CLINICAL TRIAL: NCT03856060
Title: Patient Perception of Physician's Compassion, Communication Skills, and Professionalism During Clinic Visits: a Randomized Controlled Trial (EHR Study #2)
Brief Title: Videos and Questionnaires in Assessing Patient Perception of Physician's Compassion, Communication Skills, and Professionalism During Clinic Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-1016; NCI-2019-00508 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1016 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-02-21; First posted 2019-02-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Malignant Neoplasm; Locally Advanced Malignant Neoplasm; Malignant Neoplasm; Metastatic Malignant Neoplasm; Recurrent Malignant Neoplasm
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (questionnaires, videos) (Experimental): Patients complete questionnaires and watch a video portraying a physician using a standard EHR and then another portraying a physician using an integrated model of EHR during communication over 35 minutes.
  Interventions: Other: Questionnaire Administration; Other: Video
- Group II (video, questionnaire) (Experimental): Patients complete questionnaires and watch a video portraying a physician using an integrated model of EHR and then another portraying a physician using a standard EHR during communication over 35 minutes.
  Interventions: Other: Questionnaire Administration; Other: Video

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaires
Other: Video — Watch videos of doctor and patient interaction in different settings

SUMMARY:
This trial assesses patient perception of physician's compassion, communication skills, and professionalism during clinic visits through the use of videos and questionnaires.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare patients' perception of physicians' compassion after they watch the first scripted-video vignettes of physicians: one portraying a physician using a standard electronic health record (EHR) and the other one portraying a physician using an integrated model of EHR during communication.

SECONDARY OBJECTIVES:

I. To compare patients' perception of physicians' compassion after they watch the second scripted-video vignettes of physicians: one portraying a physician using a standard electronic health record (EHR) and the other one portraying a physician using an integrated model of EHR during communication.

II. To compare patients' perception of physicians' communication skills after they watch each scripted-video vignettes of physicians: one portraying a physician using a standard EHR and the other one portraying a physician using an integrated model of EHR during communication.

III. To compare patients' perception of physicians' professionalism after they watch each scripted-video vignettes of physicians: one portraying a physician using a standard EHR and the other one portraying a physician using an integrated model of EHR during communication.

IV. To compare patients' perception of physicians' compassion, communication skills and professionalism after they watch two scripted-video vignettes of physicians: one portraying a physician using a standard electronic health record (EHR) and the other one portraying a physician using an integrated model of EHR during communication.

V. To compare patients' preference after they watch two scripted-video vignettes of physicians sequentially: one portraying a physician using a standard EHR and the other one portraying a physician using an integrated model of EHR during communication.

VI. To examine patients' perception of EHR in healthcare delivery. VII. To establish demographic and clinical factors of patients preference for the physician.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients complete questionnaires and watch a video portraying a physician using a standard electronic health record (EHR) and then another portraying a physician using an integrated model of EHR during communication over 35 minutes.

GROUP II: Patients complete questionnaires and watch a video portraying a physician using an integrated model of EHR and then another portraying a physician using a standard EHR during communication over 35 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cancer either early disease or advanced cancer defined as locally advanced, recurrent or metastatic disease.
* Outpatients (either new referrals or follow-ups) seen in the Supportive Care Clinic.
* English speaking.
* Patients with normal cognitive status (Memorial Delirium Assessment Scale [MDAS] =< 6/30) who can understand the nature and purpose of the study and have the ability to complete the consent process.

Exclusion Criteria:

* Patients who are experiencing severe symptom distress, including severe emotional distress and cognitive dysfunction, which may interfere with study participation. This will be measured by the Edmonton Symptom Assessment Scale (ESAS) and Memorial Delirium Assessment Scale (MDAS), and will be determined by the principal investigator and/or attending physician who is caring for the patient during that visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Patients' perception of physicians' compassion after they watch the first video | 1 year" or "up to 24 weeks", "through study completion
  Quantified by the total score of ratings from a comprehensive 5-item tool which assesses dimensions such as warm/cold, pleasant/unpleasant, compassionate/distant, sensitive/insensitive, and caring/uncaring (ranging from 0 to 10 for each item, and from 0 to 50 for the total score). Physicians' compassion, communication skills and professionalism will be compared between standard electronic health record (EHR) and integrated EHR groups at the end of each video using a two-sample t-test or Wilcoxon rank-sum test when appropriate. The mixed model will be applied to further explore the patterns of physicians' compassion, communication skills and professionalism from both videos. Patients' preference of physician and perception of EHR will be compared between standard EHR and integrated EHR groups using Chi-squared test or Fisher's exact test when appropriate. Logistic regression model will also be employed.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Haider, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org